CLINICAL TRIAL: NCT05890144
Title: Reconciling Relationships - An RCT Examining Relational and Clinical Decision-Making Impacts of Intensive, Brief and Control Indigenous Cultural Safety Training Interventions for Health Care Providers
Brief Title: RCT of Intensive, Brief, and Control Indigenous Cultural Safety Training Interventions for Health Care Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: St. Michael's Hospital Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RR-2019
Record Dates: First submitted 2023-05-12; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Education
Keywords: Indigenous Health; Aboriginal Health; Racism; Implicit Bias; Cultural Safety; Cultural Safety Training
MeSH Terms: conditions — Racism; Bias, Implicit

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants were not informed of the unannounced Indigenous standardized patient (UISP) visit and thus blinded to this primary outcome measure. UISPs, research and site team members were blinded to participants' study arm allocation with the exception of the study coordinator, who facilitated enrollment in intervention and control training groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intensive Intervention ("Big Canoe") (Experimental): 20 participants will be randomly assigned to Arm 1. Participants in Arm 1 ("the Big Canoe") will complete an intensive, multi-modular Indigenous cultural safety education training program that is offered online and led by trained facilitators. The curriculum in Arm 1 was developed by the San'yas Indigenous Cultural Safety Training Program in British Columbia with the support of the Ontario Indigenous Cultural Safety Training Program.
  Interventions: Other: Big Canoe
- Brief Intervention ("Little Canoe") (Active Comparator): 20 participants will be randomly assigned to Arm 2. Participants in Arm 2 ("the Little Canoe") will complete a brief, 2-hour, interactive, computer-based Indigenous race-bias education session that is offered in a computer lab with a researcher present and followed up with 2 reinforcement/reminder emails that ask questions about strategy usage at 6 and 8 weeks after the session. The intervention in Arm 2 is an Indigenous adaption of the Devine et al. (2012) anti-bias habit-breaking intervention.
  Interventions: Other: Little Canoe
- Control (Other): 20 participants will be randomly assigned to Arm 3. Participants in Arm 3 (control) will complete a primary care-related training program that is time-attention matched to Arm 1 but does not contain any content on anti-bias, anti-oppression, Indigenous peoples, or any content related to the unannounced Indigenous standardized patient encounter.
  Interventions: Other: Control

INTERVENTIONS:
Other: Big Canoe — The Big Canoe will involve an intensive, multi-modular Indigenous cultural safety education training program that is offered online and led by trained facilitators. It is 10 modules long and takes 10 weeks to complete (1 hour of learning per week).
  Arms: Intensive Intervention ("Big Canoe")
Other: Little Canoe — The Little Canoe involves a brief, 2-hour, interactive, computer-based Indigenous race-bias education session that is offered in a computer lab with a researcher present and followed up with 2 reinforcement/reminder emails that ask questions about strategy usage at 6 and 8 weeks after the session
  Arms: Brief Intervention ("Little Canoe")
Other: Control — The control is a primary care-related training program that is time-attention matched to Arm 1 but does not contain any content on anti-bias, anti-oppression, Indigenous peoples, or any content related to the unannounced Indigenous standardized patient encounter.
  Arms: Control

SUMMARY:
Despite Canada's relative global affluence, striking Indigenous/non-Indigenous health disparities persist. Following the release of the Truth and Reconciliation Commission of Canada's Final Report, and the publication of the First Peoples, Second Class Treatment report, there has been a growing recognition that the Canadian healthcare system - and the healthcare professional (HCP) - Indigenous patient relationship in particular - is a critical, necessary, and promising juncture for intervention. There has been a significant increase in the number of Indigenous cultural safety trainings for HCP across Canada. However, these programs have yet to be systematically evaluated.

This study will use a randomized parallel group design to understand and compare the effects of an intensive multi-modular Indigenous cultural safety training program (Arm 1); a brief, 2-hour, computer-based training session plus 2 follow-up emails (Arm 2); and primary care-related training program (Arm 3, control) for staff physicians, nurse practitioners, and resident physicians affiliated at large urban academic teaching hospitals in Toronto, Canada. 60 participants will be recruited and randomized into one of the three study arms. Participants will complete a series of surveys and questionnaires at baseline and 9-11 weeks post-intervention that include measures of explicit and implicit race bias.

We predict that the educational intervention in Arm 1 will have the most positive effect, followed by Arm 2 and 3 respectively. We anticipate that the results of this study will help urban hospitals implement Indigenous cultural safety training programs that are beneficial to their staff and ultimately improve the quality of care provided to Indigenous patients across Canada.

DETAILED DESCRIPTION:
STUDY PURPOSE AND OBJECTIVES

The purpose of this non-commercial, social equity, randomized control trial is to respond to the Calls for Action of the TRC by contributing to the evidence regarding the effectiveness of intensive and brief Indigenous cultural safety training programming for HCP.

The primary objective of this study is:

1. To understand and compare the relational and clinical decision-making impacts of an intensive multi-modular Indigenous cultural safety educational intervention; a brief 2-hour Indigenous race-bias educational intervention; and control intervention (primary care training that is time-attention matched to the intensive intervention) for staff physicians, resident physicians, and nurse practitioners affiliated with a large urban academic teaching hospital in Canada (St. Michael's Hospital).

The secondary objectives of this study are:

1. To document Indigenous race preference bias and differential decision making among physicians, resident physicians, and nurse practitioners affiliated with SMH.
2. To further develop and pilot Indigenous race bias educational evaluation tools and methods including a novel Indigenous Peoples in Canada - Implicit Association Test (IPC-IAT) and Indigenous Standardized Patients.
3. To build on and enhance existing San'yas and Ontario Indigenous Cultural Safety Indigenous Race Bias Training Curriculum for Health Care Providers including new modules.

STUDY DESIGN

This study is a randomized parallel group design. Participants will be randomized into one of three study arms. Participants in Arm 1 ("the Big Canoe") will complete an intensive, multi-modular Indigenous cultural safety education training program that is offered online and led by trained facilitators. The curriculum in Arm 1 was developed by study partners at the San'yas Indigenous Cultural Safety Training Program in British Columbia with the support of the Ontario Indigenous Cultural Safety Training Program. Participants in Arm 2 ("the Little Canoe") will complete a brief, 2-hour, interactive, computer-based Indigenous race-bias education session that is offered in a computer lab with a researcher present and followed up with 2 reinforcement/reminder emails that ask questions about strategy usage at 6 and 8 weeks after the session. The intervention in Arm 2 is an Indigenized version of an anti-bias education intervention developed and validated by Drs. Devine and Cox from the University of Wisconsin-Madison. Participants in Arm 3 (control) will complete a primary care-related training program that is time-attention matched to Arm 1 but does not contain any content on anti-bias, anti-oppression, Indigenous peoples, or any content related to the unannounced Indigenous standardized patient encounter. It will be administered via the Audio Digest Foundation (http://www.audio-digest.org/) platform, which houses accredited online courses for physicians and nurse practitioners.

The study proposes the use of deception practices (a temporary waiver of consent), as per Article 3.7A & B of the Tri-Council Policy Statement: Ethical Conduct for Research Involving Humans (TCPS-2).17 Each participant will be visited once by an unannounced Indigenous standardized patient (UISP) at 6-8 weeks post-intervention. The UISP will be trained to evaluate the participant's relational skills as well as their adherence to clinical guidelines. The rationale for the use of deception in this study is provided under Participant Recruitment, Enrollment, and Randomization.

STUDY SAMPLE AND SAMPLE SIZE

Participants in this study will include non-Indigenous physicians, nurse practitioners, and residents recruited from Emergency Department (ED) and the Academic Family Health Team at St. Michael's Hospital.

We aim to recruit 60 participants in each study arm, for a total of 180 participants. This should allow us to detect a difference of just under 6% in relational and clinical decision-making impact scores between treatment arms, with 20% participant attrition. This should be sufficient to, at minimum, demonstrate impact of our two intervention arms compared to control for our two primary outcomes (unannounced Indigenous standardized patient (UISP) provider relational assessment and clinical decision-making during UISP encounter).

PARTICIPANT RECRUITMENT, ENROLLMENT, AND RANDOMIZATION

Together, with each department head, Dr. Janet Smylie will provide an information session at a department staff meeting. The Research Coordinator will work with department heads to identify an appropriate departmental staff member to send an email to all of the physicians, residents, and nurse practitioners in their department that contains the study's promotional materials. The promotional materials will also be displayed in each department with the permission of the department heads. Interested staff members will be instructed in the promotional materials to contact the Research Coordinator via email or phone to learn more about the study

The Research Coordinator will be responsible for answering questions about the study and keeping track of all SMH staff who express interest in the study in an Excel spreadsheet. The Research Coordinator will email and/or hand-deliver the study information letter to SMH staff who are interested in the study. Interested staff will be instructed to visit the secure Qualtrics webpage, which will house the screening questionnaire and the study information letter and consent form. The study information letter includes information about the study purpose, procedures, risks, benefits, and measures taken to protect privacy and confidentiality.

The study proposes the use of deception as per Article 3.7 A & B of the TCPS-217, altering the requirements for consent as set out in Articles 3.1-3.5. The study proposes that each participant be visited once by an unannounced Indigenous standardized patient (UISP) at 6-8 weeks post-intervention. The UISP will be trained to evaluate the participant's relational skills as well as their adherence to clinical guidelines. The study proposes a temporary waiver of consent where participants will not be informed of the UISP visit until data collection is complete, at which time each participant will be debriefed and explicitly offered the option of refusing consent and/or withdrawing data in accordance with Article 3.7B of the TCPS2.

Immediately following completion of data collection, and prior to any analysis and/or dissemination activities, all participants will be debriefed in person by a member of the SMH research team. Debrief will be based on the findings from the UISP evaluations and not the actual recordings in order to reduce the risk of harm to the participant (i.e. personal guilt and/or incrimination). Following debrief, the SMH research team member will also explicitly offer participants the opportunity to refuse consent and/or withdraw data in accordance with Article 3.7B of the TCPS2. In addition, those individuals who have not yet completed the "Big Canoe" educational intervention will be provided the opportunity to do so, in order to ensure that all participants have fair and equal access to cultural safety training.

After consent has been obtained, participants will be prompted to enter their email to be immediately randomized into one of the study arms and to be assigned a Participant ID# . After randomization, all participants will receive an email with a link to the baseline questionnaire. This questionnaire must be completed before they begin their intervention. Participants in Arm 1, 2 and 3 will be given a link to access the online training intervention they have been randomized to receive.

Participants can withdraw from the study at any time. Participants who withdraw will not qualify for the Mainpro+ or Maintenance of Certification credits associated with the educational intervention, in its stead, they will be given the opportunity to complete the intensive online training (also accredited), for free, once the study has been completed.

DATA COLLECTION & ANALYSIS

Questionnaires At baseline, all participants will complete the following questionnaires: socio-demographic questionnaire, measures of explicit bias, the Indigenous Implicit Association Test (measure of implicit bias), and for Arm 1 only, the San'yas questionnaire. Participants will complete the same questionnaires (with the exception of the socio-demographics questionnaire) at 9-11 weeks post-intervention as well.

Unannounced Indigenous Standardized Patients Participants will also be visited by one (1) UISP without previous knowledge 8-10 weeks post-intervention completion . Indigenous actors will be hired and trained to act out a specific scenario as a UISP. Following each encounter, the UISP will complete the UISP Adherence to Clinical Practice Guidelines and UISP Cultural Safety Assessment Scoring Tool.

Data Analysis The data collected from the baseline and post-intervention questionnaires and the Indigenous standardized patients will be analyzed using the appropriate software and statistical techniques.

COMMUNITY ADVISORY BOARD

To ensure that this study does not have any negative consequences for Indigenous patients and the Indigenous communities served by St. Michael's Hospital, we have asked that the St. Michael's Hospital Indigenous Community Advisory Panel (CAP) serve as the Community Advisory Board for this trial. The Indigenous CAP has agreed to serve as the Community Advisory Board.

DISSEMINATION

The results of this study will be presented at conferences, in publications, and other public academic forums.

ELIGIBILITY:
Inclusion Criteria:

* Physicians, resident physicians, or nurse practitioners
* Non-Indigenous
* Affiliated with St. Michael's Hospital in Toronto, Canada
* Work in the Department of Family Medicine or the Emergency Department from January 2018 until 3 months post completion of training

Exclusion Criteria:

* Completion of Ontario Indigenous Cultural Safety Program or San'yas Indigenous Cultural Safety Training Program;
* Indigenous
* Intend to leave St. Michaels Hospital before 3 month post-intervention window

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Whether or not participant would be recommended as a health care provider to family or friends? | 8-10 weeks post-intervention/control
  Unannounced Standardized patient answers categorical question: "Would you recommend this health care provider to family and friends?" 4 point Likert scale (1. not recommend; 2. recommend with reservations; 3. recommend; 4. highly recommend. Higher score means better outcome
Mean Quality of Health Care Provider Relationship and Communication Scale Score | 8-10 weeks post-intervention/control
  Unannounced Indigenous Standardized patients will assess their experience of provider engagement, communication, and Indigenous cultural safety skills using the newly developed Quality of Health Care Provider Relationship and Communication Scale. Min value: 1 Max value: 5 Higher score means better outcome.
Mean Adherence to Clinical Standards of Care Scale Score | 8-10 weeks post-intervention/control
  Unannounced Indigenous Standardized patients will assess adherence of participants to clinical standards of care using developed Adherence to Clinical Standards of Care Scale for NSAID renewal and pain assessment. UISPs to present with acute flare of known ankylosing spondylitis and request NSAID renewal. History of episodic retrosternal chest pain suspicious for NSAID induced gastro-esophageal reflux disease only elicited with a review of the GI side effects of NSAIDS. Min value: 0 Max value: 22 Higher score means better outcome.

SECONDARY OUTCOMES:
Indigenous Implicit Association Test (IAT) Scores | At baseline and 9-11 weeks post-intervention/control
  The newly developed Indigenous Implicit Association Test (IAT) measures unconscious/implicit anti-Indigenous/pro-white race preference bias. Minimum score -2.0, maximum score 2.0; positive values denote a preference for white features, negative values denote a preference for Indigenous features.
Modern Prejudice Attitudes Towards Aboriginals Scale (M-PATAS) | At baseline and 9-11 weeks post-intervention/control
  14 questions and scored on a 6-point Likert scale, minimum score 1; maximum score 6; lower scores denote less prejudice; higher scores denote more prejudice
Internal Motivation to Respond Without Prejudice Scale (IMS) | At baseline and 9-11 weeks post-intervention/control
  5 questions scored on a 9-point Likert scale; Minimum score 1, Maximum score 9; higher scores denoting more internal motivation
External Motivation to Respond Without Prejudice Scale (EMS) | At baseline and 9-11 weeks post-intervention/control
  5 questions scored on a 9-point Likert scale; Minimum score 1, Maximum score 9; higher scores denoting more external motivation

CONTACTS AND LOCATIONS:
Overall Officials: Janet Smylie, MD, MPH, Principal Investigator — Well Living House, St. Michael's Hospital
Locations (1):
- Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brian Sinclair Working Group. Out of Sight. 2017. Accessed from: http://ignoredtodeathmanitoba.ca/index.php/2017/09/15/out-of-sight-interim-report-of-the-sinclair-working-group/
- [Background] Truth and Reconciliation Canada. Honouring the truth, reconciling for the future: summary of the final report of the Truth and reconciliation Commission of Canada. Winnipeg: Truth and Reconciliation Commission of Canada. 2015
- [Background] Allan, B. & Smylie, J. First Peoples, second class treatment: The role of racism in the health and well-being of Indigenous peoples in Canada. Toronto, ON: The Wellesley Institute. 2015
- [Background] Devine PG, Forscher PS, Austin AJ, Cox WT. Long-term reduction in implicit race bias: A prejudice habit-breaking intervention. J Exp Soc Psychol. 2012 Nov;48(6):1267-1278. doi: 10.1016/j.jesp.2012.06.003. PMID 23524616
- [Background] Morrison MA, Morrison TG, Harriman RL, Jewell LM. Old-fashioned and modern prejudice towards Aboriginals in Canada. In book: The Psychology of Modern Prejudice, (Ed): Morrison Melanie A., Morrison Todd G., Nova Science Publishers., Inc. 2015 pp.277-305.
- [Derived] Smylie J, Rotondi MA, Filipenko S, Cox WTL, Smylie D, Ward C, Klopfer K, Lofters AK, O'Neill B, Graham M, Weber L, Damji AN, Devine PG, Collins J, Hardy BJ. Randomized controlled trial demonstrates novel tools to assess patient outcomes of Indigenous cultural safety training. BMC Med. 2024 Jan 9;22(1):3. doi: 10.1186/s12916-023-03193-y. PMID 38191406